CLINICAL TRIAL: NCT01251237
Title: Open Study to Assess the Tolerability, Safety and Efficacy of an Adapted 2 Litre Gut Cleansing Solution (NRL0706) in Routine Colon Cleansing Prior to Colonoscopies for Colon Tumour Screening.
Brief Title: Study to Assess the Tolerability, Safety and Efficacy of an Adapted Gut Cleansing Solution in Routine Colon Cleansing Prior to Colonoscopies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Vice President, Clinical Development, Norgine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NRL0706-01/2009 (VOM); 2009-014845-95 (EudraCT Number)
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Moviprep Orange (Experimental): All patients receive 2 litres of NRL0706 solution.
  Interventions: Drug: NRL0706

INTERVENTIONS:
Drug: NRL0706 — Patients receive 1 litre of NRL0706 solution followed by 0.5 litre of clear liquid during the afternoon/evening prior to colonoscopy. Patients receive 1 litre of 0706 solution followed by 0.5 litre of clear liquid during the morning of colonoscopy.

SUMMARY:
It is particularly important that thorough gut cleansing is achieved prior to the colonoscopy for the procedure to be successful. Polyethylene glycol plus electrolyte (PEG+E) solutions are well established as safe and effective agents for gut cleansing and Norgine has successfully developed a low volume (2 litre) PEG+E gut lavage solution. The efficacy and safety of this solution is similar to the standard 4 litre PEG+E, but with improved patient acceptance.

Tolerance, acceptability and satisfaction with the cleansing agent plays an important role in subjects' compliance with gut preparation procedure. The study medication NRL0706 is identical to the PEG+E-containing gut lavage solution commonly used in clinical practice, with the exception that the flavour has been modified from lemon to orange. This study is to investigate the tolerability, acceptability, safety and efficacy of a single dose of NRL0706 (MOVIPREP Orange) in subjects without gastrointestinal symptoms undergoing colonoscopy for colon cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* The subject's written informed consent must be obtained prior to inclusion.
* Male or female ambulatory subjects aged between 40 to 75 years undergoing a complete colonoscopy for colon cancer screening.
* No history of significant gastrointestinal diseases, including gastrointestinal obstruction and perforation or acute symptoms requiring a colonoscopy procedure.
* Willing to undergo a colonoscopy for colon cancer screening.
* Willing, able and competent to complete the entire procedure and to comply with study instructions.
* Females of childbearing potential must employ an adequate method of contraception.

Exclusion Criteria:

* History of gastric emptying disorders
* History of ileus, toxic megacolon, gastrointestinal obstruction and colonic perforation
* History of Phenylketonuria
* Known Glucose-6-phosphate dehydrogenase deficiency
* Known hypersensitivity to macrogol 3350, sodium sulphate or ascorbic acid/ sodium ascorbate
* History of colonic resection
* Requirement for permanent medication and associated stable serum concentrations (e.g. neuroleptic drugs)
* Presence of congestive heart failure (NYHA III + IV)
* Acute life-threatening cardiovascular disease
* Documented history of severe renal insufficiency
* Application of any unlicensed medication within the previous 3 months or participation in any other research study in the last 3 months
* Females who are pregnant, nursing or planning a pregnancy. Females of child bearing potential not using reliable methods of contraception
* Subjects who the investigator feels would not be compliant with the requirements of the trial

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Overall Acceptance on VAS (100mm) rating | 12 hours

SECONDARY OUTCOMES:
Tolerance on five-point VRS | 12 hours
Taste Evaluation on VAS (100mm) rating | 12 hours
Acceptability rated by compliance, four-point VRS and VAS (100mm) rating | 12 hours
Efficacy on five-grade scale for pre-defined colon areas | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Fischbach, Prof Dr med, Principal Investigator — Klinikum Aschaffenburg-Alzenau
Locations (1):
- Wolfgang Fischback, Aschaffenburg, Germany